CLINICAL TRIAL: NCT04482582
Title: Early Percutaneous Cryoablation for Pain Control After Rib Fractures Among Elderly Patients
Acronym: EPERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Joseph Forrester, Assistant Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 57099
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08

CONDITIONS: Rib Fractures
Keywords: rib fractures, CT guided cryoneurolysis
MeSH Terms: conditions — Rib Fractures | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: We are proposing a prospective, randomized trial evaluating efficacy of image-guided percutaneous intercostal cryoneurolysis (pICN) for pain control after traumatic rib fractures in persons >=65 years. Eligible patients would be enrolled by the trauma service after consent or assent is obtained. Patients will be randomized to either pICN within 72 hours of presentation or existing standard-of-care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Image-guided percutaneous ICN (pICN): Group A (Experimental): Patients who were admitted after a traumatic injury, with rib fractures identified, who are >= 65 years of age will be randomized to percutaneous image-guided cryoneurolysis (pICN) group within 72 hours of presentation.
  Interventions: Radiation: Cryoneurolysis
- Standard-of Care : Group B (Active Comparator): Patients who were admitted after a traumatic injury, with rib fractures identified, who are >= 65 years of age will be randomized to standard-of-care group within 72 hours of presentation.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Radiation: Cryoneurolysis — Patients will be offered a minimally invasive solution known as cryoneurolysis. By directly applying a cold cryoneurolysis probe to the nerves the axon is destroyed, resulting in Wallerian degeneration of the distal nerve without distorting epineurial or perineurial tissue. Application of cryoneurolysis will help reduce the amount of narcotics the patient would need to take and instead provide them longer term pain control with minimal risk.
  Arms: Image-guided percutaneous ICN (pICN): Group A
Other: Standard of Care — Patients will be provided regular standard of care at the Stanford Hospital with long-term follow-up provided at the Stanford Center for Reconstruction after Chest Wall Injury.
  Arms: Standard-of Care : Group B

SUMMARY:
The purpose of this study is to provide long-term pain control for elderly patients with rib fractures in order to minimize their risk of complications and return them to baseline functional capacity

DETAILED DESCRIPTION:
The purpose of this study is to provide long-term pain control for elderly patients with rib fractures in order to minimize their risk of complications and return them to baseline functional capacity. In order to do this, we would offer a minimally invasive solution known as Cryoneurolysis. By directly applying cold Cryoneurolysis to the nerves, this can destroy nerve axons, resulting in Wallerian degeneration of the distal nerve without distorting epineural or perineurial tissue. The application of cryoneurolysis will help reduce the amount of narcotics the patient would need, and potentially lead to a better post-injury quality of life.

ELIGIBILITY:
Inclusion criteria:

i) Patients greater than 65 years with any acute rib fracture

ii) Pain score equal to or greater than 5 with deep inspiration.

iii) Presenting and admitted to Stanford Emergency Department

Exclusion criteria:

i) Radiographic evidence of metastasis to ribs

ii) Glasgow Coma Scale (GCS) score <13

iii) Patients undergoing SSRF

iv) Rib fractures located < 3cm from spinous process

v) Coagulopathy (INR >1.5, Pat < 100)

vi) Other factors precluding cryoablation at IR attending's discretion

vii) If only ribs broken are 1,2 or 10,11, 12

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Acute Pain Assessed by Numeric Pain Score | Hospital discharge (up to 1 month)
  The patient will be asked to verbalize their numeric pain score daily after hospital discharge. Pain measured on a scale of 0 to 10, with 0 being no pain and 10 being the worst pain.
  Note: The timing of hospital discharge varies by patient as these are polytrauma patients.

SECONDARY OUTCOMES:
30-day mortality | 1 month after hospital discharge
  Will be obtained from chart review after discharge
Number of participants requiring ICU admission | 1 month after hospital discharge
  Will be obtained from chart review after discharge
Length of hospital stay | Up to 1 month
  The Length of Stay will be obtained from the patient's chart after discharge and will depend on the level of care required for recovery from their injuries.
Use of Narcotic Equivalents | Hospital discharge (up to 1 month), 1 month, 3 months, 12 months after hospital discharge
  Daily oral narcotic equivalents
30-day rib-specific readmission | 1 month after hospital discharge
  Incidence of readmission. The patient will be admitted back to the hospital if pain level relates to rib-specific injuries such as hemothorax and pneumonia.
The McGill Pain Questionnaire (MPQ) and Pain Rating Index (PRI) Scale Score | 1 month, 3 months, 12 months (all from hospital discharge)
  The McGill Pain Questionnaire (MPQ) is a validated 20 question instrument to quantify subjective pain and the scoring system yields a Pain Rating Index (PRI) score between Mild, Moderate or Severe. The questionnaire will be administered to the patient by study/ clinical staff upon discharge. The scoring system yields a pain rating index (PRI) score between 0 and 50 used to temporally track pain, higher scores correspond to higher pain levels.
The Glasgow Outcome Scale Extended (GOS-E) Score | 1 month, 3 months, 12 months (all from hospital discharge)
  The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories: Dead, Vegetative State, Severe Disability, Moderate Disability or Good Recovery. The Extended GOS (GOSE) provides more detailed categorization into eight categories by subdividing the categories of severe disability, moderate disability and good recovery into a lower and upper category:
  1. Death (D)
  2. Vegetative state (VS)
  3. Lower severe disability (SD -)
  4. Upper severe disability (SD +)
  5. Lower moderate disability ( MD -)
  6. Upper moderate disability ( MD +)
  7. Lower good recovery (GR -)
  8. Upper good recovery (GR +)
  The questionnaire will be administered to the patient by study/clinical staff upon discharge.
Short Form (SF-12) Health Survey Scale Score | 1 month, 3 months, 12 months (all from hospital discharge)
  The 12-Item Short-Form Health Survey is a widely used composite score used to gauge overall health. The composite score is based on 8 domains scores contained in the SF-12 questionnaire, which will be administered to the patient by study/clinical staff upon discharge.
  Score ranges from 1 (Excellent) to 5 (Poor) , 1 (Yes, limited a lot) to 3 (No, not limited at all), 1 (Yes) 2 (No), 1 (Not at all) to 5 (Extremely), 1 (All of the time) to 6 (None of the time) and 1 (All of the time) to 5 (None of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Forrester, MD, Principal Investigator — Stanford University; Nishita Kothary, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Sharma OP, Oswanski MF, Jolly S, Lauer SK, Dressel R, Stombaugh HA. Perils of rib fractures. Am Surg. 2008 Apr;74(4):310-4. doi: 10.1177/000313480807400406. PMID 18453294
- [Background] Marasco S, Lee G, Summerhayes R, Fitzgerald M, Bailey M. Quality of life after major trauma with multiple rib fractures. Injury. 2015 Jan;46(1):61-5. doi: 10.1016/j.injury.2014.06.014. Epub 2014 Jun 21. PMID 25069400
- [Background] Fabricant L, Ham B, Mullins R, Mayberry J. Prolonged pain and disability are common after rib fractures. Am J Surg. 2013 May;205(5):511-5; discusssion 515-6. doi: 10.1016/j.amjsurg.2012.12.007. PMID 23592156
- [Background] Gordy S, Fabricant L, Ham B, Mullins R, Mayberry J. The contribution of rib fractures to chronic pain and disability. Am J Surg. 2014 May;207(5):659-62; discussion 662-3. doi: 10.1016/j.amjsurg.2013.12.012. Epub 2014 Jan 31. PMID 24612969
- [Background] Holcomb JB, McMullin NR, Kozar RA, Lygas MH, Moore FA. Morbidity from rib fractures increases after age 45. J Am Coll Surg. 2003 Apr;196(4):549-55. doi: 10.1016/S1072-7515(02)01894-X. PMID 12691929
- [Background] Stawicki SP, Grossman MD, Hoey BA, Miller DL, Reed JF 3rd. Rib fractures in the elderly: a marker of injury severity. J Am Geriatr Soc. 2004 May;52(5):805-8. doi: 10.1111/j.1532-5415.2004.52223.x. PMID 15086666
- [Background] Bulger EM, Arneson MA, Mock CN, Jurkovich GJ. Rib fractures in the elderly. J Trauma. 2000 Jun;48(6):1040-6; discussion 1046-7. doi: 10.1097/00005373-200006000-00007. PMID 10866248
- [Background] Liman ST, Kuzucu A, Tastepe AI, Ulasan GN, Topcu S. Chest injury due to blunt trauma. Eur J Cardiothorac Surg. 2003 Mar;23(3):374-8. doi: 10.1016/s1010-7940(02)00813-8. PMID 12614809
- [Background] Van Vledder MG, Kwakernaak V, Hagenaars T, Van Lieshout EMM, Verhofstad MHJ; South West Netherlands Trauma Region Study Group. Patterns of injury and outcomes in the elderly patient with rib fractures: a multicenter observational study. Eur J Trauma Emerg Surg. 2019 Aug;45(4):575-583. doi: 10.1007/s00068-018-0969-9. Epub 2018 Jun 15. PMID 29905897
- [Background] Witt CE, Bulger EM. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. Trauma Surg Acute Care Open. 2017 Jan 5;2(1):e000064. doi: 10.1136/tsaco-2016-000064. eCollection 2017. PMID 29766081
- [Background] Todd SR, McNally MM, Holcomb JB, Kozar RA, Kao LS, Gonzalez EA, Cocanour CS, Vercruysse GA, Lygas MH, Brasseaux BK, Moore FA. A multidisciplinary clinical pathway decreases rib fracture-associated infectious morbidity and mortality in high-risk trauma patients. Am J Surg. 2006 Dec;192(6):806-11. doi: 10.1016/j.amjsurg.2006.08.048. PMID 17161098
- [Background] de Jong MB, Kokke MC, Hietbrink F, Leenen LP. Surgical Management of Rib Fractures: Strategies and Literature Review. Scand J Surg. 2014 Jun;103(2):120-125. doi: 10.1177/1457496914531928. Epub 2014 Apr 29. PMID 24782038
- [Background] Shi HH, Esquivel M, Staudenmayer KL, Spain DA. Effects of mechanism of injury and patient age on outcomes in geriatric rib fracture patients. Trauma Surg Acute Care Open. 2017 Mar 16;2(1):e000074. doi: 10.1136/tsaco-2016-000074. eCollection 2017. PMID 29766084
- [Background] Tignanelli CJ, Rix A, Napolitano LM, Hemmila MR, Ma S, Kummerfeld E. Association Between Adherence to Evidence-Based Practices for Treatment of Patients With Traumatic Rib Fractures and Mortality Rates Among US Trauma Centers. JAMA Netw Open. 2020 Mar 2;3(3):e201316. doi: 10.1001/jamanetworkopen.2020.1316. PMID 32215632
- [Background] Pieracci FM, Majercik S, Ali-Osman F, Ang D, Doben A, Edwards JG, French B, Gasparri M, Marasco S, Minshall C, Sarani B, Tisol W, VanBoerum DH, White TW. Consensus statement: Surgical stabilization of rib fractures rib fracture colloquium clinical practice guidelines. Injury. 2017 Feb;48(2):307-321. doi: 10.1016/j.injury.2016.11.026. Epub 2016 Nov 27. No abstract available. PMID 27912931
- [Background] Chen Zhu R, de Roulet A, Ogami T, Khariton K. Rib fixation in geriatric trauma: Mortality benefits for the most vulnerable patients. J Trauma Acute Care Surg. 2020 Jul;89(1):103-110. doi: 10.1097/TA.0000000000002666. PMID 32176172
- [Background] Kulminski AM, Ukraintseva SV, Kulminskaya IV, Arbeev KG, Land K, Yashin AI. Cumulative deficits better characterize susceptibility to death in elderly people than phenotypic frailty: lessons from the Cardiovascular Health Study. J Am Geriatr Soc. 2008 May;56(5):898-903. doi: 10.1111/j.1532-5415.2008.01656.x. Epub 2008 Mar 21. PMID 18363679
- [Background] Farhat JS, Velanovich V, Falvo AJ, Horst HM, Swartz A, Patton JH Jr, Rubinfeld IS. Are the frail destined to fail? Frailty index as predictor of surgical morbidity and mortality in the elderly. J Trauma Acute Care Surg. 2012 Jun;72(6):1526-30; discussion 1530-1. doi: 10.1097/TA.0b013e3182542fab. PMID 22695416
- [Background] Abellan van Kan G, Rolland Y, Houles M, Gillette-Guyonnet S, Soto M, Vellas B. The assessment of frailty in older adults. Clin Geriatr Med. 2010 May;26(2):275-86. doi: 10.1016/j.cger.2010.02.002. PMID 20497846
- [Background] Ryb GE, Dischinger PC, Burch CA, Kerns TJ, Kufera J, Andersen D. Frailty and injury causation. Ann Adv Automot Med. 2012;56:175-81. PMID 23169127
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Background] Ilfeld BM. Continuous Peripheral Nerve Blocks: An Update of the Published Evidence and Comparison With Novel, Alternative Analgesic Modalities. Anesth Analg. 2017 Jan;124(1):308-335. doi: 10.1213/ANE.0000000000001581. PMID 27749354
- [Background] Janssen TL, Hosseinzoi E, Vos DI, Veen EJ, Mulder PGH, van der Holst AM, van der Laan L. The importance of increased awareness for delirium in elderly patients with rib fractures after blunt chest wall trauma: a retrospective cohort study on risk factors and outcomes. BMC Emerg Med. 2019 Jun 13;19(1):34. doi: 10.1186/s12873-019-0248-z. PMID 31195982
- [Background] Ilfeld BM, Preciado J, Trescot AM. Novel cryoneurolysis device for the treatment of sensory and motor peripheral nerves. Expert Rev Med Devices. 2016 Aug;13(8):713-25. doi: 10.1080/17434440.2016.1204229. Epub 2016 Jul 13. PMID 27333989
- [Background] Keller BA, Kabagambe SK, Becker JC, Chen YJ, Goodman LF, Clark-Wronski JM, Furukawa K, Stark RA, Rahm AL, Hirose S, Raff GW. Intercostal nerve cryoablation versus thoracic epidural catheters for postoperative analgesia following pectus excavatum repair: Preliminary outcomes in twenty-six cryoablation patients. J Pediatr Surg. 2016 Dec;51(12):2033-2038. doi: 10.1016/j.jpedsurg.2016.09.034. Epub 2016 Sep 28. PMID 27745867
- [Background] Harbaugh CM, Johnson KN, Kein CE, Jarboe MD, Hirschl RB, Geiger JD, Gadepalli SK. Comparing outcomes with thoracic epidural and intercostal nerve cryoablation after Nuss procedure. J Surg Res. 2018 Nov;231:217-223. doi: 10.1016/j.jss.2018.05.048. Epub 2018 Jun 21. PMID 30278932
- [Background] Vossler JD, Zhao FZ. Intercostal nerve cryoablation for control of traumatic rib fracture pain: A case report. Trauma Case Rep. 2019 Jul 31;23:100229. doi: 10.1016/j.tcr.2019.100229. eCollection 2019 Oct. PMID 31388539
- [Background] Koethe Y, Mannes AJ, Wood BJ. Image-guided nerve cryoablation for post-thoracotomy pain syndrome. Cardiovasc Intervent Radiol. 2014 Jun;37(3):843-6. doi: 10.1007/s00270-013-0718-8. Epub 2013 Aug 17. PMID 23954965
- [Background] Byas-Smith MG, Gulati A. Ultrasound-guided intercostal nerve cryoablation. Anesth Analg. 2006 Oct;103(4):1033-5. doi: 10.1213/01.ane.0000237290.68166.c2. PMID 17000825
- [Background] Pieracci FM, Leasia K, Bauman Z, Eriksson EA, Lottenberg L, Majercik S, Powell L, Sarani B, Semon G, Thomas B, Zhao F, Dyke C, Doben AR. A multicenter, prospective, controlled clinical trial of surgical stabilization of rib fractures in patients with severe, nonflail fracture patterns (Chest Wall Injury Society NONFLAIL). J Trauma Acute Care Surg. 2020 Feb;88(2):249-257. doi: 10.1097/TA.0000000000002559. PMID 31804414
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Marasco SF, Martin K, Niggemeyer L, Summerhayes R, Fitzgerald M, Bailey M. Impact of rib fixation on quality of life after major trauma with multiple rib fractures. Injury. 2019 Jan;50(1):119-124. doi: 10.1016/j.injury.2018.11.005. Epub 2018 Nov 3. PMID 30442372
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Derived] Liou RJ, Earley MJ, Forrester JD. Effect of climate on surgical site infections and anticipated increases in the United States. Sci Rep. 2022 Nov 16;12(1):19698. doi: 10.1038/s41598-022-24255-w. PMID 36385136